CLINICAL TRIAL: NCT04981405
Title: Real-world Evidence of COVID-19 Vaccine Effectiveness Against COVID-19 Hospitalization: the Case-control Study in St. Petersburg, Russia
Brief Title: Real-world Evidence of COVID-19 Vaccines Effectiveness
Status: Terminated | Type: Observational
Why Stopped: low recruitment, end of COVID-19 pandemic
Sponsor: Ivan S Moiseev (Other)
Collaborators: European University at St. Petersburg (Other); Medical Institute named after Berezin Sergey (Unknown)
Responsible Party: Sponsor-Investigator, Ivan S Moiseev, Dr, St. Petersburg State Pavlov Medical University
Organization: St. Petersburg State Pavlov Medical University (Other)
Other Study IDs: CDRU-003
Record Dates: First submitted 2021-07-26; First posted 2021-07-29 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients hospitalised to clinics of First Pavlov State Medical University of Saint - Petersburg: 450 cases - patients hospitalised with COVID-19 450 control - patients hospitalised without COVID-19 in the same period (surgical, oncological, cardiological, ophthalmologic, gastroenterological departments)
  Interventions: Biological: COVID-19 Vaccines
- Patients referred to Medical Institute named after Berezin Sergey for computed tomography: Cases - patients with pneumonia confirmed after computed tomography. Controls - patients without pneumonia after computed tomography.
  Interventions: Biological: COVID-19 Vaccines

INTERVENTIONS:
Biological: COVID-19 Vaccines — "Gam-COVID-Vac" "EpiVacCorona" "COVIVAC"

SUMMARY:
This is an observational case-control study to evaluate COVID-19 vaccine effectiveness against hospitalisation with COVID-19 related conditions in St. Petersburg, Russia. Two sets of cases and control will be retrospectively analyzed to compare vaccination proportions and other characteristics to infer vaccine effectiveness from odds ratios. The first set of cases will be extracted from the data on hospitalisation of patients with COVID-19 to First Pavlov State Medical University of Saint-Petersburg hospitals, and controls will be patients hospitalised with other conditions. The second set of cases and controls will be based on patients referred to Medical Institute named after Berezin Sergey for computed tomography. Cases will be patients with positive SARS-CoV-2 status computed tomography confirmed pneumonia or patients referred to hospitalisation, and control will be patients without pneumonia and not referred to hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized to clinics of First Pavlov State Medical University of Saint-Petersburg
* Patients referred to Medical Institute named after Berezin Sergey for computed tomography
* Available vaccination status

Exclusion Criteria:

- Refusal to provide information for research purposes at the time of hospitalization or reference to computed tomography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of Saint-Petersburg, Russia
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Effectiveness of full vaccination against hospitalization with COVID-19 pneumonia | 3 months
  Full vaccination effectiveness is calculated based on the odds ratio of vaccination proportions in cases and controls, adjusted for other patient characteristics. Full vaccination status is assigned after two weeks of the second dose for each vaccine separately.

SECONDARY OUTCOMES:
Effectiveness of partial vaccination against hospitalization with COVID-19 pneumonia | 3 months
  Partial vaccination effectiveness is calculated based on the odds ratio of vaccination proportions in cases and controls, adjusted for other patient characteristics. Partial vaccination status is assigned after two weeks of the first dose for each vaccine separately.
Effectiveness of vaccination against hospitalization with COVID-19 pneumonia in different age groups | 3 months
  Evaluate vaccine effectiveness in different age groups (<20, 20-29, 30-39, 40-49, 50-59, 60-69, >70)

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Mikhail Cherkashin, Saint Petersburg, Sankt-Peterburg
  - Oksana Stanevich, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Barchuk A, Bulina A, Cherkashin M, Berezina N, Rakova T, Kuplevatskaya D, Skougarevskiy D, Okhotin A. Gam-COVID-Vac, EpiVacCorona, and CoviVac effectiveness against lung injury during Delta and Omicron variant surges in St. Petersburg, Russia: a test-negative case-control study. Respir Res. 2022 Oct 10;23(1):276. doi: 10.1186/s12931-022-02206-3. PMID 36217139